CLINICAL TRIAL: NCT05107544
Title: Metabolic, Physical Fitness and Mental Health Effects of High Intensity Interval Training (HIIT) in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Las Higueras (Other)
Collaborators: Hospital Guillermo Grant Benavente (Unknown); Centro de Vida Saludable, Universidad de Concepción (Unknown)
Responsible Party: Principal Investigator, JULIO SOTO BARROS, Pediatric endocrinologist, Hospital Las Higueras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-12-67
Record Dates: First submitted 2021-10-11; First posted 2021-11-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Interval Training (Experimental): The entire group is going to be undergo the intervention
  Interventions: Other: HIGH INTENSITY INTERVAL TRAINING

INTERVENTIONS:
Other: HIGH INTENSITY INTERVAL TRAINING — Will be prescribed HIIT through online modality to a group of adolescents with type 1 diabetes 3 times a week for 3 months. The training is going to have 2 phases, the initial phase and improvement phase, which are going to be differentiated according to work intensity following the recommendations of the American College of Sports Medicine. During the initial phase (first 4 weeks) the intensity is going to be 60-75% of the VO2 max. During the improvement phase the intensity is going to increase to a 75-85% of the VO2 max for 8 week.

SUMMARY:
Patients with type 1 diabetes usually present cardiovascular risk factors. Sixty percent of them are overweight or obese, 40% have hypertension, 60% have dyslipidemia, leading to cardiovascular disease as the major cause of death in adults with type 1 diabetes. Regular exercise can help patients to improve cardiovascular disease risk profile, metabolic control and chronic complications. Recommendations for exercise in children with diabetes are the same as the general population, between ages 8 to 18 years 60 min of physical exercise/day is suggested, including moderate or vigorous aerobic activity (at least 20 minutes), muscle strengthening and bone strengthening activities. Children with type 1 diabetes have poorer physical fitness levels than the non-diabetic peers and it has been described some barriers to meet these recommendations between children and adolescents with type 1 diabetes such as the fear of hypoglycemia, external temperature, work schedule, loss of control of diabetes, a low fitness level. The two types of exercise (aerobic and anaerobic) are recommended in people with diabetes. High intensity interval training involves alternation between brief periods of vigorous exercise and recovery at low to moderate intensity. Has been shown that HIIT is associated with improving aerobic capacity without a detrimental decline in blood glucose in adults with type 1 diabetes and home-based high-intensity interval training reduces barriers to exercise in the same group. The objective of the present study is to propose a HIIT exercise protocol through online modality to a group of adolescents with type 1 diabetes to evaluate the metabolic effects and physical capacity through an analytical, prospective and longitudinal study (before and after) for 3 months. As primary outcome is expected to improve metabolic control shown as an increase in time in range on continuous glucose monitoring and a decrease in glycosylated hemoglobin. And as secondary results, improve the aerobic capacity and resistance strength, lipid profile parameters, anthropometric and on the mood of the participants.

DETAILED DESCRIPTION:
Hypothesis Three month HIIT training program increases time in range (TIR) and decreases glycemic variability (MAGE) in adolescents with DM1.

HIIT training program improves physical fitness (aerobic capacity and strength) of adolescents with DM1.

Methodology Analytical, prospective, longitudinal study (before and after). This type of study was chosen for ethical reasons. A group will not be left without intervention knowing the benefits of physical exercise in patients with DM1.

HIIT for 3 months

Population of study This study will be carried out with adolescents with type 1 diabetes treated at the sponsoring Hospitals: Las Higueras and Guillermo Grant Benavente.

A sample size of 30 Adolescents would be sufficient to detect a 15 percent increase in the percentage of time in the range of glucose values within the target range four months after the study start using a level of significance of 0.05% a power of 80% and a loss of follow-up of 15% (4 adolescents).

Type of sampling Convenience sampling

Procedures

Metabolic control monitoring Continuous glucose monitoring (CGM) will be used continuously during the study period. The duration of the CGM is going to be 7 days each time (Guardian Connect, Medtronic). If the patients are already wearing a CGM, will use the same device and data from these specific times will be collected for analysis.

Blood glucose will be monitored during exercise to make adjustments to therapy if necessary. This will be done by the doctors weekly for the first month and then every 15 days.

The statistical analysis of the continuous glucose monitoring (CGM) will be carried out in 4 moments: before starting the study, the first month after, at 3 months and 3 months after ending the training.

Blood sampling is going to be taken at baseline and at 3 month. will be measured HbA1c and lipid profile.

Total insulin dosing is going to be carefully recorded as units/kg/day during the study.

An insulin sensitivity score (ISS) is going to be calculated using the SEARCH ISS model: logeIS = 4.64725 - 0.02032 × (waist, cm) - 0.09779 × (HbA1c, %) - 0.00235 × (TG, mg/dL; R2 = 0.74 in the initial SEARCH model). This has been validated using the hyperinsulinemic euglycemic clamp, considered the gold standard for insulin sensitivity measures. CGM data are going to be downloaded and used to calculate percent blood glucose at, below, or above target.

The HbA1c and lipid profile will be measured using the Abbott brand model Architect c8000.

Nutritional assessment Nutritional consultation is going to be performed to the participants, in which it will be carried out a body composition analysis using the bioimpedianciometer TANITA TBF-40 at several times: before starting the intervention, at 1 month, at 3 months and at 3 months after finishing the intervention.

Two educational sessions will be performed to participants and parents and / or caregivers on carbohydrate content and glycemic index to reinforce the knowledge acquired throughout the course of the pathology in order to contribute to improve glycemic control. These will be carried out through a digital platform divided into groups of 10 or 15 participants.

In order to know the daily calorie intake and the distribution of macronutrients of the participants, the information from the 24-hour reminder questionnaire will be collected through a telephone call in 4 random days (without prior notice) during the same evaluation times mentioned previously.

Fitness monitoring Before intervention the participants are going to undergo physical evaluation: Cafra test, course-navette test, strength and Physical activity questionnaire for adolescents (PAQ-a) to determine their health-related fitness before applying the protocol. To standardize the sample and avoid cardiovascular risks due to the intensity of the effort, the Cafra test will be applied, which will enable the participant to perform the following tests. This test is used in the evaluation of physical education by the Education Quality Measurement System in the country. At the end of intervention aerobic capacity and resistance strength is going to be evaluated again.

The Cafra test goal is to determine the cardiovascular adaptive capacity of the participants from workloads of medium intensity during walking. If at the end of the test the individual has a heart rate equal to or greater than 160 beats per minute, he should not take the Navette test.

The Navette test is a cardiorespiratory fitness test. The moment in which the individual interrupts the test indicates the cardiorespiratory endurance. In addition, at the time this test is performed, blood pressure will be measured before and at the end, to rule out the presence of baseline or exercise-induced hypertension.

The heart rate will be measured with a heart rate sensor, which indicates in real time the heart rate reached, during the initial and final evaluations and during training sessions.

To evaluate muscular endurance, the abdominal test will be performed in 60 seconds and the largest possible number of push-ups without rest will be carried out. In this way, there will be a record of how the physical condition is before and after applying the protocol.

Adherence to physical training and nutritional consultations will be monitored through the online connection.

Physical training The training is going to have 2 phases, the initial phase and improvement phase, which are going to be differentiated according to work intensity following the recommendations of the American College of Sports Medicine. To prescribe the intensity of exercise karvonen formula is going to be used for which resting heart rate measured for a week is needed.

The methodology of work is going to be High intensity interval training (HIIT) using cardiovascular and endurance exercises using the own weight considering an intensity of 60-75% of the VO2max during the first 4 weeks (initial phase). The frequency of the training is 3 times a week under researcher online supervision between 3 to 7 pm Monday to Friday. During the improvement phase the intensity is going to increase to a 75-85% of the VO2max for 8 week. The intensity and effects of the training will be monitored thought heart rate sensors and the Borg Rating of Perceived Exertion Scale. Post-exercise monitoring, class coordination, reminders and motivation to participate will be performed by online group administered by the researchers.

Two physical education teachers will supervise each session.

Strategies to avoid acute changes in glycemia during training

It will be required that participants check the blood glucose by fingerstick before meals, before and after exercise, at bedtime, and twice a week around midnight.

The amount and type of food are not going to be controlled, but will be asked participants not exercising before or within 90 minutes after a meal . Considering that HIIT is associated to stable glycaemia no changes will be prescribed in fast-acting insulin dose.

For the management of blood glucose levels during the training period (before, during and after each session), a protocol based on the recommendations of the consensus for glycemia management during exercise using continuous glucose monitoring will be used.

Before starting and after completing each training session, a capillary blood glucose measurement will be requested as a safety measure and also in the event of symptoms of hypoglycemia or if the sensor shows or anticipates hypoglycemia.

In addition, when participants first start exercising, according to the midnight glycemia, it may be necessary to reduce the basal insulin dose by 20-50% on the day of exercise.

Participants using an insulin pump will use the same protocol, with a reduction in bolus doses and use of temporary basal on the days of exercise.

Mood evaluation The Patient Health Questionnaire 9 (PHQ-9) will be applied in its version for adolescents, which consists of nine questions designed to evaluate depressive symptoms according to DSM-5 criteria, on an ordinal scale according to the frequency of symptoms (never, some days, more than half of the days, almost every day). The score range is from 0 to 27 points, where higher values indicate a greater probability of a Depressive Episode. This scale is graded into 4 categories: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderate to severe), 20-27 (severe). According to recent evidence, a score greater than or equal to 11 is recommended as a cut-off point to determine probable depressive episode in the Chilean population of adolescents. Patients who present a cut-off point higher than this in the initial evaluation will be excluded from protocol and will be referred to child psychiatry care.

To evaluate the effects of exercise on the depressed mood of adolescents, this survey will also be applied at the end of the intervention and 3 months after the intervention.

Blood Pressure Measurement In addition, during the initial evaluation, blood pressure will be measured before and after the physical tests to detect children with suspected hypertension, who as detailed above will be excluded from the intervention.

The BP recording will be carried out with an oscillometric device and the conditions for this procedure are: the adolescent must be seated, with the right arm uncovered, feet resting on the floor, and the BP cuff at the level of the heart. Before measuring the blood pressure the individual will need to remain sitting for at least five minutes. The blood pressure value will be evaluated according to the recommendations for the diagnosis of hypertension in children and adolescents of the American Academy of Pediatrics.

Statistical Analysis The initial analysis will examine data distribution through the Shapiro-Wilk test and baseline characteristics of all adolescents.

The quantitative variables will be expressed as means or medians, accompanied by deviation or interquartile ranges according to the exploration of normality. It will be analyzed each time of evaluation (transversal) using the chi-square test for categorical variables and the Student-t or Wilcoxon tests for continuous variables.

Relevant tests will be used to consider the non-dependence of the data obtained for both qualitative and quantitative analysis.

The effects of the treatment will be expressed , using mixed regression models (longitudinal) adjusting for potential confounders at baseline.

Subgroup analysis will be performed with interaction tests for relevant variables as BMI and socioeconomic status. Two separate definitions of compliance will be used. First, adolescents will be considered compliant to the HIIT treatment if participation is at least 75% of the number of training. Second, adolescents will be considered compliant to the HIIT if attendance is 100% of the counseling sessions to the nutritional and to endocrine consultations.

Outcome comparisons in the time will be analyzed intention-to-treat basis, regardless of whether is abandoned the study or fully adhere to the intervention. A secondary per-protocol analysis will be performed for the primary outcome including only the adolescents who were compliant with the protocol.

All analyses will follow a pre-specified statistical analysis plan. Stata v.14 software (StataCorp, College Station, TX) will be used for statistical analysis.

ELIGIBILITY:
The eligibility criteria will be applied to the group of patients treated at Las Higueras Hospital and Guillermo Grant Benavente Hospital

Inclusion Criteria:

* Adolescents with type 1 diabetes
* Ages: 12-19 years (and in pubertal stage of at least Tanner stage III breast or genitalia)
* HbA1c between 7 and 11.5%
* Total daily insulin dose ≥0.7 units/kg/day.
* Both genders
* Patients treated regularly at Las Higueras Hospital and Guillermo Grant Benavente Hospital.

Exclusion Criteria:

* < 1 year of diabetes
* Any medical, mental or physical disability that contraindicates exercise.
* Practice of regular, structured and planned physical exercise outside the project, more than 2 times a week.
* Pregnancy or breastfeeding
* > 1 episode of severe hypoglycemia in the last 6 months

Eligibility criteria:

If the patient meets the inclusion criteria and does not present exclusion criteria, he/she may proceed to carry out physical evaluations to determine if has the conditions to perform the intervention. The patient may be ineligible for investigation in case of:

* Upon completing the Cafra test, His/her heart rate is> or equal to 160 (20, 23)
* If he/she shows blood pressure compatible with arterial hypertension before or after the initial physical evaluation.

Definition of arterial hypertension according to the recommendations of the American Academy of Pediatrics (30):

Blood pressure> or equal to the 95th percentile or> 130/80 mm Hg in adolescents greater than or equal to 13 years.

* If he/she develops any signs of post-exercise musculoskeletal injury (functional impotence, pain or swelling joint)
* In case they present a score ≥11 in the PHQ-9 questionnaire without mental health evaluation.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Time change in range | First month after starting training
  Time in Range (TIR) is the percentage of time that a person spends with their blood glucose levels in a target range (70-180)
Time change in range | Three months after starting training
  Time in Range (TIR) is the percentage of time that a person spends with their blood glucose levels in a target range (70-180)
Time change in range | Three months after finishing training
  Time in Range (TIR) is the percentage of time that a person spends with their blood glucose levels in a target range (70-180)

SECONDARY OUTCOMES:
Change in hemoglobin A1c | Three months after starting training
  Blood test
Change in hemoglobin A1c | Three months after finishing training
  Blood test
Change in cholesterol | Three months after starting training
  Blood test
Change in cholesterol | Three months after finishing training
  Blood test
Change in triglycerides | Three months after starting training
  Blood test
Change in triglycerides | Three months after finishing training
  Blood test
Changes in systolic blood pressure | Three months after starting training
  Blood pressure monitor
Changes in systolic blood pressure | Three months after finishing training
  Blood pressure monitor
Changes in body composition | Three months after starting training
  The participant's weight will be taken with a calibrated scale
Changes in body composition | Three months after finishing training
  The participant's weight will be taken with a calibrated scale
Changes in body composition | Three months after starting training
  The participant's height will be taken with a tape measure
Changes in body composition | Three months after finishing training
  The participant's height will be taken with a tape measure
Changes in waist circumference | Three months after starting training
  The participant's waist circumference will be taken with a tape measure
Changes in waist circumference | Three months after finishing training
  The participant's waist circumference will be taken with a tape measure
Changes in aerobic capacity | Three months after starting training
  Will be done through the Navetta test
Changes in aerobic capacity | Three months after finishing training
  Will be done through the Navetta test
Change in heart rate | Three months after starting training
  It will be measured with a heart rate sensor, which indicates in real time the heart rate reached
Change in heart rate | Three months after finishing training
  It will be measured with a heart rate sensor, which indicates in real time the heart rate reached
Change in resistance strength | Three months after starting training
  It will be tested with repeated contractions for a period of time long enough for muscle fatigue to occur. The abdominal test will be performed in 60 seconds and the largest possible number of push-ups without rest will be performed
Change in resistance strength | Three months after finishing training
  It will be tested with repeated contractions for a period of time long enough for muscle fatigue to occur. The abdominal test will be performed in 60 seconds and the largest possible number of push-ups without rest will be performed
Change in total insulin dose | Three months after starting training
  Blood test
Change in total insulin dose | Three months after finishing training
  Blood test
Frequency of hypoglycemia episodes during the training | Three months after starting training
  A blood glucose meter will be used and trained to report episodes during workouts
Frequency of hypoglycemia episodes during the training | Three months after finishing training
  A blood glucose meter will be used and trained to report episodes during workouts
Change in mood of adolescents | Three months after starting training
  Application of the PHQ-9 questionnaire. This scale is graded into 4 categories: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderate to severe), 20-27 (severe) (25). A score greater than or equal to 11 is recommended as a cut-off point to determine probable ED in the Chilean population of adolescents
Change in mood of adolescents | Three months after finishing training
  Application of the PHQ-9 questionnaire. This scale is graded into 4 categories: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderate to severe), 20-27 (severe) (25). A score greater than or equal to 11 is recommended as a cut-off point to determine probable ED in the Chilean population of adolescents

CONTACTS AND LOCATIONS:
Overall Officials: JULIO SOTO, MD, Principal Investigator — Hospital Las Higueras
Locations (1):
- Hospital Las Higueras, Talcahuano, Concepcion, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller RG, Mahajan HD, Costacou T, Sekikawa A, Anderson SJ, Orchard TJ. A Contemporary Estimate of Total Mortality and Cardiovascular Disease Risk in Young Adults With Type 1 Diabetes: The Pittsburgh Epidemiology of Diabetes Complications Study. Diabetes Care. 2016 Dec;39(12):2296-2303. doi: 10.2337/dc16-1162. Epub 2016 Sep 21. PMID 27654986
- [Background] Riddell, M., & Perkins B. (2006). Type 1 diabetes and vigorous exercise: Applications of exercise physiology to patient management. Canadian journal of diabetes, 30(1), 63-71.
- [Background] MacMillan F, Kirk A, Mutrie N, Matthews L, Robertson K, Saunders DH. A systematic review of physical activity and sedentary behavior intervention studies in youth with type 1 diabetes: study characteristics, intervention design, and efficacy. Pediatr Diabetes. 2014 May;15(3):175-89. doi: 10.1111/pedi.12060. Epub 2013 Jul 29. PMID 23895512
- [Background] Katz M, Giani E, Laffel L. Challenges and Opportunities in the Management of Cardiovascular Risk Factors in Youth With Type 1 Diabetes: Lifestyle and Beyond. Curr Diab Rep. 2015 Dec;15(12):119. doi: 10.1007/s11892-015-0692-4. PMID 26520142
- [Background] Adolfsson P, Riddell MC, Taplin CE, Davis EA, Fournier PA, Annan F, Scaramuzza AE, Hasnani D, Hofer SE. ISPAD Clinical Practice Consensus Guidelines 2018: Exercise in children and adolescents with diabetes. Pediatr Diabetes. 2018 Oct;19 Suppl 27:205-226. doi: 10.1111/pedi.12755. No abstract available. PMID 30133095
- [Background] Kriska AM, LaPorte RE, Patrick SL, Kuller LH, Orchard TJ. The association of physical activity and diabetic complications in individuals with insulin-dependent diabetes mellitus: the Epidemiology of Diabetes Complications Study--VII. J Clin Epidemiol. 1991;44(11):1207-14. doi: 10.1016/0895-4356(91)90153-z. PMID 1941015
- [Background] Jabbour G, Henderson M, Mathieu ME. Barriers to Active Lifestyles in Children with Type 1 Diabetes. Can J Diabetes. 2016 Apr;40(2):170-2. doi: 10.1016/j.jcjd.2015.12.001. PMID 27038139
- [Background] Scott SN, Cocks M, Andrews RC, Narendran P, Purewal TS, Cuthbertson DJ, Wagenmakers AJM, Shepherd SO. High-Intensity Interval Training Improves Aerobic Capacity Without a Detrimental Decline in Blood Glucose in People With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Feb 1;104(2):604-612. doi: 10.1210/jc.2018-01309. PMID 30281094
- [Background] Scott SN, Shepherd SO, Strauss JA, Wagenmakers AJM, Cocks M. Home-based high-intensity interval training reduces barriers to exercise in people with type 1 diabetes. Exp Physiol. 2020 Apr;105(4):571-578. doi: 10.1113/EP088097. Epub 2019 Oct 25. PMID 31584734
- [Background] Reddy R, Wittenberg A, Castle JR, El Youssef J, Winters-Stone K, Gillingham M, Jacobs PG. Effect of Aerobic and Resistance Exercise on Glycemic Control in Adults With Type 1 Diabetes. Can J Diabetes. 2019 Aug;43(6):406-414.e1. doi: 10.1016/j.jcjd.2018.08.193. Epub 2018 Aug 30. PMID 30414785
- [Background] Clements MA, Foster NC, Maahs DM, Schatz DA, Olson BA, Tsalikian E, Lee JM, Burt-Solorzano CM, Tamborlane WV, Chen V, Miller KM, Beck RW; T1D Exchange Clinic Network. Hemoglobin A1c (HbA1c) changes over time among adolescent and young adult participants in the T1D exchange clinic registry. Pediatr Diabetes. 2016 Aug;17(5):327-36. doi: 10.1111/pedi.12295. Epub 2015 Jul 8. PMID 26153338
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Hasan R, Perez-Santiago D, Churilla JR, Montes B, Hossain J, Mauras N, Darmaun D. Can Short Bouts of Exercise ("Exercise Snacks") Improve Body Composition in Adolescents with Type 1 Diabetes? A Feasibility Study. Horm Res Paediatr. 2019;92(4):245-253. doi: 10.1159/000505328. Epub 2020 Jan 31. PMID 32007996
- [Background] Quirk H, Blake H, Dee B, Glazebrook C. "You can't just jump on a bike and go": a qualitative study exploring parents' perceptions of physical activity in children with type 1 diabetes. BMC Pediatr. 2014 Dec 20;14:313. doi: 10.1186/s12887-014-0313-4. PMID 25526774
- [Background] Francois ME, Baldi JC, Manning PJ, Lucas SJ, Hawley JA, Williams MJ, Cotter JD. 'Exercise snacks' before meals: a novel strategy to improve glycaemic control in individuals with insulin resistance. Diabetologia. 2014 Jul;57(7):1437-45. doi: 10.1007/s00125-014-3244-6. Epub 2014 May 10. PMID 24817675
- [Background] Mauras N, Beck R, Xing D, Ruedy K, Buckingham B, Tansey M, White NH, Weinzimer SA, Tamborlane W, Kollman C; Diabetes Research in Children Network (DirecNet) Study Group. A randomized clinical trial to assess the efficacy and safety of real-time continuous glucose monitoring in the management of type 1 diabetes in young children aged 4 to <10 years. Diabetes Care. 2012 Feb;35(2):204-10. doi: 10.2337/dc11-1746. Epub 2011 Dec 30. PMID 22210571
- [Background] Dabelea D, D'Agostino RB Jr, Mason CC, West N, Hamman RF, Mayer-Davis EJ, Maahs D, Klingensmith G, Knowler WC, Nadeau K. Development, validation and use of an insulin sensitivity score in youths with diabetes: the SEARCH for Diabetes in Youth study. Diabetologia. 2011 Jan;54(1):78-86. doi: 10.1007/s00125-010-1911-9. Epub 2010 Oct 1. PMID 20886205
- [Background] American College of Sports Medicine (2014). Manual ACSM para la valoración del fitness relacionado con la salud. España: Wolters Kluwer Health.
- [Background] American College of Sports Medicine. (2007). Manual ACSM para la valoración y prescripción del ejercicio. Madrid, España: Paidotribo.
- [Background] Shepherd SO, Wilson OJ, Taylor AS, Thogersen-Ntoumani C, Adlan AM, Wagenmakers AJ, Shaw CS. Low-Volume High-Intensity Interval Training in a Gym Setting Improves Cardio-Metabolic and Psychological Health. PLoS One. 2015 Sep 24;10(9):e0139056. doi: 10.1371/journal.pone.0139056. eCollection 2015. PMID 26402859
- [Background] Shepherd SO, Cocks M, Tipton KD, Ranasinghe AM, Barker TA, Burniston JG, Wagenmakers AJ, Shaw CS. Sprint interval and traditional endurance training increase net intramuscular triglyceride breakdown and expression of perilipin 2 and 5. J Physiol. 2013 Feb 1;591(3):657-75. doi: 10.1113/jphysiol.2012.240952. Epub 2012 Nov 5. PMID 23129790
- [Background] Tsalikian E, Mauras N, Beck RW, Tamborlane WV, Janz KF, Chase HP, Wysocki T, Weinzimer SA, Buckingham BA, Kollman C, Xing D, Ruedy KJ; Diabetes Research In Children Network Direcnet Study Group. Impact of exercise on overnight glycemic control in children with type 1 diabetes mellitus. J Pediatr. 2005 Oct;147(4):528-34. doi: 10.1016/j.jpeds.2005.04.065. PMID 16227041
- [Background] Riddell MC, Scott SN, Fournier PA, Colberg SR, Gallen IW, Moser O, Stettler C, Yardley JE, Zaharieva DP, Adolfsson P, Bracken RM. The competitive athlete with type 1 diabetes. Diabetologia. 2020 Aug;63(8):1475-1490. doi: 10.1007/s00125-020-05183-8. Epub 2020 Jun 12. PMID 32533229
- [Background] Scott SN, Shepherd SO, Andrews RC, Narendran P, Purewal TS, Kinnafick F, Cuthbertson DJ, Atkinson-Goulding S, Noon T, Wagenmakers AJM, Cocks M. A Multidisciplinary Evaluation of a Virtually Supervised Home-Based High-Intensity Interval Training Intervention in People With Type 1 Diabetes. Diabetes Care. 2019 Dec;42(12):2330-2333. doi: 10.2337/dc19-0871. Epub 2019 Sep 17. PMID 31530660
- [Background] Lee AS, Johnson NA, McGill MJ, Overland J, Luo C, Baker CJ, Martinez-Huenchullan S, Wong J, Flack JR, Twigg SM. Effect of High-Intensity Interval Training on Glycemic Control in Adults With Type 1 Diabetes and Overweight or Obesity: A Randomized Controlled Trial With Partial Crossover. Diabetes Care. 2020 Sep;43(9):2281-2288. doi: 10.2337/dc20-0342. Epub 2020 Jul 9. PMID 32647051
- [Background] Campos Jara C, Delgado Floody P, Caamano Navarrete F, Guzman Guzman I, Cesp Barria M, Jerez Mayorga D, Alarcon Hormazabal M, Osorio Poblete A. Alteraciones en el rendimiento fisico de escolares: los Test Cafra y Navette y su asociacion con la obesidad y riesgo cardiometabolico. Nutr Hosp. 2016 Jul 19;33(4):374. doi: 10.20960/nh.374. Spanish. PMID 27571652
- [Background] Huerta Ojeda A, Galdames Maliqueo S, Cataldo Guerra M, Barahona Fuentes G, Rozas Villanueva T, Caceres Serrano P. [Effects of a high intensity interval training on the aerobic capacity of adolescents]. Rev Med Chil. 2017 Aug;145(8):972-979. doi: 10.4067/s0034-98872017000800972. Spanish. PMID 29189854
- [Background] Agencia de calidad de la educación. (2018). Informe de resultados estudio nacional, Educación física 8° básico. Recuperado de https://archivos.agenciaeducacion.cl/Informe_de_Resultados_Estudio_Nacional_Educacion_Fisica_8_Basico_2018.pdf
- [Result] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459